CLINICAL TRIAL: NCT05833776
Title: Value of IPACK Block (Interspace Between the Popliteal Artery and Capsule of Knee) With Spinal Anesthesia Versus Fentanyl Based Spinal Anesthesia on Postoperative Analgesia for Knee Arthroscopic Meniscectomy
Brief Title: Value of IPACK Block (Interspace Between the Popliteal Artery and Capsule of Knee) With Spinal Anesthesia Versus Fentanyl Based Spinal Anesthesia for Knee Arthroscopic Meniscectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, mohamed A Aboelsuod, MD, assistant professor of anesthesia intensive care and pain management, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 91945931
Record Dates: First submitted 2023-04-05; First posted 2023-04-27 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Post Operative Pain
Keywords: IPACK Block, spinal anesthesia, Knee arthroscopy.
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group F (Experimental): received spinal anesthesia using hyperbaric bupivacaine 0.5% (3ml) with fentanyl (25ug)
  Interventions: Procedure: spinal anesthesia using hyperbaric bupivacaine 0.5% (3ml) with fentanyl (25ug)
- group I (Experimental): group I (30 patients) received spinal anesthesia using hyperbaric bupivacaine 0.5% (3ml) with IPACK Block using plain bupivacaine 0.5% (15ml).
  Interventions: Procedure: spinal anesthesia using hyperbaric bupivacaine 0.5% (3ml) with fentanyl (25ug)

INTERVENTIONS:
Procedure: spinal anesthesia using hyperbaric bupivacaine 0.5% (3ml) with fentanyl (25ug) — group I (30 patients) received spinal anesthesia using hyperbaric bupivacaine 0.5% (3ml) with IPACK Block using plain bupivacaine 0.5% (15ml).

SUMMARY:
Postoperative analgesia is provided by local anesthesia combined with intrathecal narcotics. In addition, for the first 24 hours, this combination has a parenteral opioid sparing effect. However, despite its benefits, this method has been associated to an increased incidence of urine retention, nausea, and vomiting, as well as pruritus. A new localized analgesic approach called as IPACK (infiltration between the knee capsule and the popliteal artery) has been employed in practice.

DETAILED DESCRIPTION:
The goal of this study was to compare fentanyl based spinal anesthesia to IPACK Block-based spinal anesthesia during knee arthroscopy.

Patients and Methods: The study enrolled sixty patients with ASA (I-II) ranging in age from 25 to 60 years old after receiving ethical committee permission and written informed consent from patients. They were divided into two groups: group F (30 patients) received spinal anesthesia using hyperbaric bupivacaine 0.5% (3ml) with fentanyl (25ug) and group I (30 patients) received spinal anesthesia using hyperbaric bupivacaine 0.5% (3ml) with IPACK Block using plain bupivacaine 0.5% (15ml). Results: In the first 4 hours postoperatively, there were no variations in VAS scores between the two groups; however, following 4 hours and over the next 12 hours, Group I, VAS scores were lower. The amount of morphine used overall was lower in Group I, which took longer than Group F to reach initial rescue analgesia. The level of patient satisfaction 48 hours after surgery was higher in group I than in group F.

ELIGIBILITY:
Inclusion Criteria:

age from 25 to 60 years old, with ASA physical status I-III undergoing for knee arthroscopy

Exclusion Criteria:

Patient refusal, neuromuscular diseases, allergies to local anesthetics, and contraindications to spinal anesthesia such as coagulopathy and severe mitral stenosis

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
post-operative analgesia | 24 hours
  post-operative pain relief

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No